CLINICAL TRIAL: NCT03209050
Title: Evaluation of the Surfacer System Approach to Central Venous Access
Acronym: SAVEUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merit Medical Systems, Inc. (Industry)
Collaborators: Meditrial Europe Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BVT.Surfacer.17-01
Record Dates: First submitted 2017-06-16; First posted 2017-07-06 (Actual); Results first posted 2021-08-12 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Venous Occlusion

STUDY DESIGN:
Intervention Model Description: patients requiring venous access
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Central Venous Access Placement (Other): Central venous access placement
  Interventions: Device: Central Venous Access Placement

INTERVENTIONS:
Device: Central Venous Access Placement — Device inserted into the femoral vein to insert a central venous access catheter

SUMMARY:
Pre-market Investigational device exemption study evaluating the safety and efficacy of the Surfacer System to facilitate stable upper body central venous access suitable for any conventional catheter.

DETAILED DESCRIPTION:
This prospective, single arm, multi-center study is to demonstrate the safety and efficacy of the Surfacer System. Safety will be evaluated based on the overall rate of acute complications using the study device as compared to historical rates of device/procedure related safety events using conventional central venous access methods. Efficacy will be evaluated by the rate of transient successful central venous accesses created by the study device. A total of 30 patients are planned to be enrolled, with 10 patients initially following review of safety data. Duration expected to be through 7 days. A minimum of 3 sites will participate in the study in the United States.

ELIGIBILITY:
Inclusion Criteria:

* referred for placement of central venous access catheter
* have limited or diminishing upper body venous access
* have pathology impeding standard access methods
* willing to give written informed consent

Exclusion Criteria:

* occlusion of the right femoral vein
* occlusion of the iliac vein
* occlusion of the inferior vena cava
* contraindicated by physician
* acute thrombosis within any vessel planned to be crossed by the Surfacer *tortuous anatomy which precludes a straight line from femoral vein to subclavian
* diagnosed with active pericarditis
* diagnosed with active endocarditis
* suspected pericardial effusion
* known or suspected aneurysm or ectasia of ascending aorta
* innominate artery or subclavian artery
* pregnant or of childbearing potential not taking adequate contraceptive measures or nursing during study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Tocchi, MD, Study Director — Meditrial Europe Ltd.
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Central Venous Access Placement
Started | 30
Completed | 27
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: patients with central venous disease with pathology impeding standard access methods
Arm/Group | Central Venous Access Placement
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants] | 30
Region of Enrollment [Number; unit: participants]
  United States | 30
chronic Kidney disease [Count of Participants; unit: Participants] | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Safe Insertion and Patency of Central Venous Access Catheter
Description: Safety reported as 86.7% (26/30) % of subjects with no procedural complications at discharge through 7 days follow up.
Time Frame: 7 days
Measure: Number; unit: participants
Groups:
- Central Venous Access Placement: Central venous access placement in 26/30 patients
  Central Venous Access Placement: Device inserted into the femoral vein to insert a central venous access catheter in 26/30 patients
Arm/Group | Central Venous Access Placement
Number analyzed (Participants) | 30
participants | 30
Statistical Analysis 1: Comparison: Central Venous Access Placement; Test type: Other; p = 0.5, Clopper-Pearson 95% CI

2. Secondary Outcome: Number of Participants Who Experienced Safe Use of the System to Insert Femoral Vein to Sub-clavicular Exit as Assessed by Central Venous Access Placement in 30 Patients Attempted
Description: Safety and Efficacy 90.0% (27/30) successful central venous catheter placements as assessed by patent open central venous access catheter. Ability to use the central venous access catheter for dialysis and infusion through 7 days
Time Frame: 7 days
Population: patients treated with central venous access device
Measure: Count of Participants; unit: Participants
Groups:
- Central Venous Access Placement: Central venous access placement in 27/30 patients
  Central Venous Access Placement: Device inserted into the femoral vein to insert a central venous access catheter in 27/30 patients
Arm/Group | Central Venous Access Placement
Number analyzed (Participants) | 30
Participants | 30

ADVERSE EVENTS:
Time Frame: 4 weeks or 30 days
Description: Overall number of participants who experienced adverse events as a result of the access procedure per definitions within 24 hours of occurrence.
Arm/Group | Central Venous Access Placement
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 4/30
Other Adverse Events (participants affected / at risk) | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Central Venous Access Placement (N=30)
Hypotension (Renal and urinary disorders) | 1 (1) — Hypovolemia causing Hypotension post dialysis, resolved with inpatient hospitalization greater than 24 hours
Bleeding (Vascular disorders) | 2 (2) — Bleeding requiring transfusion and narcan and colloidal solution. In patient hospitalization greater than 24 hours
Hemodynamic Instability (Vascular disorders) | 1 (1) — low blood pressure requiring vasopressors, extended hospitalization greater than 24 hours
unintended embolization (Vascular disorders) | 1 (1) — anticoagulants administered, in patient hospitalization greater than 24 hours
bleeding (Vascular disorders) | 2 (2) — bleeding at the central venous access site, resolved with transfusion
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Central Venous Access Placement (N=30)
allergic reaction (Infections and infestations) | 1 (1) — one allergic reaction occurred rated as mild adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT03209050/Prot_SAP_000.pdf